CLINICAL TRIAL: NCT05801536
Title: The Effects of Transcutaneous Electrical Stimulation on Arm Functions in Individuals With Cervical Spinal Cord Injury.
Brief Title: TCES for Upper Limb Function in Cervical SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: International Spinal Research Trust (Other)
Responsible Party: Principal Investigator, Professor Sarah Astill, Associate Professor in Motor Control, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMN007
Record Dates: First submitted 2023-03-16; First posted 2023-04-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries
Keywords: transcutaneous electrical stimulation; cervical; upper limbs
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper limb task practice with or without cervical transcutaneous electrical stimulation (Experimental): Task specific practice will be combined with cervical transcutaneous electrical stimulation.
  Interventions: Device: SCONE

INTERVENTIONS:
Device: SCONE — This is a noninvasive (nonsurgical) electrical neuromodulation device to reactivate and retrain the neurons and neural networks in the spinal cord to improve function after neurological trauma. The device will be used to stimulate the cervical spinal cord as participants practice tasks involving upper limb control.

SUMMARY:
Following a cervical spinal cord injury (cSCI; damage to the spinal cord at the neck) there is catastrophic loss of hand and grip function. This has a devastating effect on quality of life and functional independence. Thus, there is a real need to identify and optimise therapy to aid functional arm and hand recovery. One such therapy is Transcutaneous Electrical Stimulation (tCES). This involves applying sticky pads to the skin and then transmitting a low-level electrical current to the spinal cord. This activates neural circuits, allowing injured nerves to transmit signals to muscles to produce movement while completing upper limb tasks. The purpose of this pilot project is to establish if and how tCES might be used to improve arm and hand control. The investigators will recruit 8 people who have had a cSCI for >1yr. First, the investigators will invite volunteers to the University for 2 weeks, twice per week, to establish their baseline movement capacity.

Then the investigators will allocate the volunteers to one of two groups: group 1 will undertake 4 weeks of upper limb task practice (ULTP) followed by 4 weeks of ULTP+tCES; group 2 will undertake ULTP+tCES for 4 weeks followed by 4 weeks of ULTP. Participants will then complete a week (2 sessions) of post-intervention assessment. The investigators will then invite volunteers and carers to be interviewed about their experiences of being involved in the project. Finally, there will be 2 sessions of follow-up assessment after 3 months. In order to assess if and how ULTP+tCES affects arm and hand control the investigators will measure: movement capacity using standard clinical tests; muscular activity in response to brain/spinal stimulation; how fast and smooth movements are when reaching and grasping objects. The investigators will also examine how the intervention has affected Quality of Life (QoL) and independence (Spinal Cord Independence Measure).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) can be defined as a loss of communication between the brain and the body due to damage to pathways within the spinal cord. Injury to the cervical levels of the spinal cord are more common than injury to the lower segments of the spinal cord, thus tetraplegia is more common than paraplegia (Thompson et al., 2014). Tetraplegics rank regaining arm and hand function as their main priority for rehabilitation, five times greater than bowel, bladder, sexual or lower extremity function (Anderson, 2004). However, compared to recent advances made in recovery of ambulatory function, research that strives to uncover how best to optimise arm/hand rehabilitation after SCI is very limited. Thus identifying and optimising efficacious therapies to restore functional arm and hand recovery is an important clinical, economic and social goal.

While promising molecular strategies have emerged to reduce secondary injury and promote axonal regrowth, an effective cure eludes people with cervical SCI, and overall recovery of arm and hand function using these means remains limited (Levi et al., 2018). Functional training, or task specific training of a motor function (e.g. reaching and grasping), is currently the most effective evidence-based way of enhancing plasticity to recover motor function. A promising approach is the use of stimulation-based rehabilitative therapies promoting neural plasticity along the spinal cord/corticospinal tract. Among these, transcutaneous electrical stimulation (TCES) (Gerasimenko et al., 2015) was demonstrated to be effective for improving hand grip strength in people with spinal cord injury (Gad et al., 2018). The investigators hypothesise that combining upper limb practice (ULTP) and TCES to the cervical spinal cord over the course of 4 weeks, could affect arm/ hand function and quality of life to a greater extent than ULTP by itself.

The principal aim of the study is to test the effects of transcutaneous electrical stimulation on arm and hand functions in individuals with cervical spinal cord injury. In addition, the investigators aim to assess the neurophysiological mechanisms with which transcutaneous electrical stimulation supports the observed changes in hand/arm function.

The primary objective of the study is to measure and compare the changes in hand and arm functions, assessed through the Graded and Redefined Assessment of Strength, Sensibility and Prehension test (GRASSP) tool, occurring over the course of the two interventions (ULTP and ULTP + TCES). In addition, secondary objectives are:

To explain the neurophysiological mechanisms with which transcutaneous electrical stimulation results in changes in hand/arm function.

To establish a clearly defined, reproducible protocol for establishing participant specific TCES settings.

To understand factors that contribute to participants wanting to use TCES and their experience of using TCES.

The study will consist of two weeks of baseline measurements, 8 weeks of intervention (4 weeks of ULTP and 4 weeks of TCES + ULTP) in a cross-over design, followed by two-weekly and a 3 month follow-up with no further intervention (Inanici et al., 2018). The baseline measurements (see primary and secondary outcome measures) are necessary to document stability of functional status. Baseline measures will take place over 2 sessions, each week (e.g. 4 baseline testing sessions).

Participation to the study will span over the course of 25 weeks. On the first 2 weeks, participants will attend the lab twice per week. On the following 8 weeks, participants will attend the lab three times per week. On week 11, participants will attend the lab twice. On week 12, participants and their carers will be invited to a semi-structured interview. There will then be a 3-months break during which the participants are not required to attend the lab, after which (week 25) they will take part on two follow-up sessions.

ELIGIBILITY:
Inclusion Criteria:

Cervical (between C3 and C7) spinal cord injury at least 1 year prior to the study.

* Between 18 and 80 years of age.
* Difficulty with hand functions in activities of daily living (e.g. dressing, grooming, feeding)
* Stable medical condition without cardiopulmonary disease or frequent autonomic dysreflexia that would contraindicate participation in upper extremity rehabilitation or testing activities.
* Capable of performing simple cued motor tasks such as reaching and touching or grasping objects.
* Ability to attend 3 sessions of weekly experimental sessions and testing activities over the course of 8 weeks.
* Ability to provide informed consent (either verbally or in writing).
* Ability to read/speak English.

Exclusion Criteria:

* History of additional neurologic disease, such as stroke, multiple sclerosis, traumatic brain injury, etc.
* Peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.).
* Rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.).
* Active cancer
* Cardiovascular or pulmonary disease that would prevent full participation in the upper limb practice intervention
* Ongoing medical complications (such as unhealed fracture, contracture, pressure sore, or urinary tract infection or other illnesses) that might interfere with upper extremity rehabilitation or testing activities
* Any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician
* Personal or familial history of epilepsy
* Pregnancy
* Botulinum toxin injections in the prior 6 months
* Dependent on ventilation support
* Implanted stimulator (e.g. vagus nerve stimulator, pacemaker, cochlear implant, etc) 0r infusion device (e.g. insulin pump, etc).
* Cardiac pacemaker or intracardial lines. Exclusions for general safety
* Pregnancy
* Alcohol and/or drug abuse.
* Unable to read and/or comprehend the consent form.
* Unable to understand the instructions given as part of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
GRASSP | 17 months
  Graded and Redefined Assessment of Strength, Sensibility and Prehension test. The primary objective of the study is to measure and compare the changes in hand and arm functions, assessed through the Graded and Redefined Assessment of Strength, Sensibility and Prehension test (GRASSP) tool, occurring over the course of the two interventions (ULTP and ULTP + TCES).

SECONDARY OUTCOMES:
Kinematics movement time | 17 months
  The time (seconds) taken to complete the reach to grasp tasks
Kinematics peak velocity | 17 months
  The maximum velocity (m/s) value observed during the reach to grasp tasks
Surface Electromyography (sEMG) amplitude | 17 months
  The root mean square amplitude (rms) of EMG signals during unimanual and bimanual standardised reach to grasp actions will be monitored.
Surface Electromyography (sEMG) frequency | 17 months
  The frequency (Hz) of EMG signals during unimanual and bimanual standardised reach to grasp actions will be monitored.
Spinal-evoked potentials | 17 months
  Upon electrical stimulation at the cervical level spinally evoked potentials in forearm muscles including biceps brachii (biceps), triceps brachii (triceps), extensor carpi radialis (ECR), flexor carpi radialis (FCR) and abductor pollicis brevis (APB) will be investigated.
Motor Evoked Potentials | 17 months
  Motor-evoked potentials recorded from the dominant (APB) muscle induced via transcranial magnetic stimulation will be monitored.
Monosynaptic reflex | 17 months
  Evoked upon median nerve stimulation in FCR and APB muscles.
Spinal Cord Independence Measure (SCIM) questionnaire score | 17 months
  Measures independence across 3 sub-domains. Range 0 to 100 with 100 indicating better independence
Quality of Life (QoL) questionnaire score. | 17 months
  Measures quality of life according to measures of satisfaction and importance across multiple domains. Scale 1-6 with 6 indicating more satisfied or more important

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Astill, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No